CLINICAL TRIAL: NCT05386147
Title: Pilot Study to Observe Effects of Flourish HEC Vaginal Care System on Vaginal Microbiome in Women With Recurrent Bacterial Vaginosis
Brief Title: Flourish HEC to Prevent Recurrence of BV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vaginal Biome Science (Other)
Collaborators: Center for Pelvic Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BV2P0821
Record Dates: First submitted 2022-05-11; First posted 2022-05-23 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Bacterial Vaginosis
Keywords: BV recurrence; probiotic; intravaginal gel; vaginal pH; vulvovaginal symptoms questionnaire
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: A single group of women with recurrent bacterial vaginosis who elect to participate in the study will be assessed before and after using a vaginal care system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study group (Experimental): Women with recurrent BV use the Flourish HEC Vaginal Care System, consisting of three components: 1) "Balance" external wash; 2) BioNourish vaginal moisturizing gel (an FDA 510k cleared class II medical device); and 3) BiopHresh homeopathic vaginal suppository with probiotics. All system components are currently available to the public at national retailers. Women will use the system for six months. They will have vaginal microbiome composition (next-generation sequencing and Nugent score) and vaginal pH tested at baseline, 3 months, and 6 months. At each timepoint they will also complete the vulvovaginal symptoms questionnaire (VSQ).
  Interventions: Device: Flourish HEC Vaginal Care System (contains a class II medical device plus other unregulated components)

INTERVENTIONS:
Device: Flourish HEC Vaginal Care System (contains a class II medical device plus other unregulated components) — see arm description

SUMMARY:
In a population of women with heightened vulvovaginal sensitivity and recurrent bacterial vaginosis (BV), the use of the Flourish HEC Vaginal Care System is being tested for prevention of BV recurrence over six months of use.

DETAILED DESCRIPTION:
BV treated with metronidazole or clindamycin recurs within 3 months in at least 43% of women, requiring additional rounds of antibiotics. Preliminary data show that the use of a commercially available 3-component kit can dramatically reduce BV recurrence over 11 weeks of use. This study tests a similar kit with one component altered - the intravaginal gel is composed of hydroxyethylcellulose rather than aloe, making it less likely to trigger reactions in women with sensitive tissues. The study will examine recurrence of BV, vaginal pH, and vulvovaginal symptoms as in the prior study, though extended to 6 months. Additionally, this study examines changes in the vaginal microbiome using targeted next-generation sequencing with the use of the Flourish HEC system.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women between the ages of 18 and 52.
* Diagnosis of recurrent BV: >= 3 episodes of BV within last year, or >= 2 episodes of BV within past six months, recorded in medical record
* Desire to use personal hygiene products to avoid recurrence of BV.

Exclusion Criteria:

* Known allergy or sensitivity to any other ingredient in the Flourish HEC Vaginal Care System
* Immunosuppressed or immunocompromised individuals
* Known allergy or intolerability to metronidazole
* Anyone who may have mental health disorders triggered by answering questions related to vulvar or vaginal health, by pelvic exams, or self-application of vaginal products
* Known vaginal infection that is not BV or yeast infection
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Change in vaginal microbiome by next-generation sequencing (NGS) | Baseline to 3 months
  Vaginal swab will be analyzed by commercially available NGS service
Change in vaginal microbiome by next-generation sequencing (NGS) | Baseline to 6 months
  Vaginal swab will be analyzed by commercially available NGS service
Change in vaginal microbiome by next-generation sequencing (NGS) | 3 months to 6 months
  Vaginal swab will be analyzed by commercially available NGS service
Change in vaginal microbiome by Nugent scoring | Baseline to 3 months
  Vaginal smear slide will be Gram stained and Nugent scored
Change in vaginal microbiome by Nugent scoring | Baseline to 6 months
  Vaginal smear slide will be Gram stained and Nugent scored
Change in vaginal microbiome by Nugent scoring | 3 months to 6 months
  Vaginal smear slide will be Gram stained and Nugent scored
BV recurrence | 6 months
  Percentage of women with recurrence of BV during the study after initial cure with routine care, if applicable

SECONDARY OUTCOMES:
Change in vulvovaginal symptoms questionnaire (VSQ) self-report | Baseline to 3 months
  Vaginal and vulvar symptoms will be self-reported using validated VSQ modified to 4-point Likert scores. VSQ consists of a series of questions, each of which is rated as 0 (never), 1(rarely), 2(sometimes), 3 (frequently). Lower scores are healthier. Each question is analyzed separately; there is no overall score reported.
Change in vulvovaginal symptoms questionnaire (VSQ) self-report | Baseline to 6 months
  Vaginal and vulvar symptoms will be self-reported using validated VSQ modified to 4-point Likert scores. VSQ consists of a series of questions, each of which is rated as 0 (never), 1(rarely), 2(sometimes), 3 (frequently). Lower scores are healthier. Each question is analyzed separately; there is no overall score reported.
Change in vulvovaginal symptoms questionnaire (VSQ) self-report | 3 months to 6 months
  Vaginal and vulvar symptoms will be self-reported using validated VSQ modified to 4-point Likert scores. VSQ consists of a series of questions, each of which is rated as 0 (never), 1(rarely), 2(sometimes), 3 (frequently). Lower scores are healthier. Each question is analyzed separately; there is no overall score reported.
Change in vaginal pH | Baseline to 3 months
  Vaginal pH will be tested using pH strip
Change in vaginal pH | Baseline to 6 months
  Vaginal pH will be tested using pH strip
Change in vaginal pH | 3 months to 6 months
  Vaginal pH will be tested using pH strip

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kellogg-Spadt, PhD, CRNP, Principal Investigator — Center for Pelvic Medicine
Locations (1):
- Center for Pelvic Medicine, Rosemont, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chidawanyika, Tamutenda PhD; Cathy Yi, Chung Hwa MD; Kelly-Martin, Rachel; Cleland, Joshua PhD; DuPriest, Elizabeth PhD Preliminary Data from Clinical Trial to Survey Results of Flourish Vaginal Care System for Recurrent BV [A80], Obstetrics & Gynecology: May 2022 - Volume 139 - Issue - p 24S doi: 10.1097/01.AOG.0000826648.49549.01